CLINICAL TRIAL: NCT03096457
Title: Topical Paromomycin Cream For Bolivian Cutaneous Eishmaniasis: A Controlled Study
Brief Title: Topical Paromomycin for Cutaneous Leishmaniasis in Bolivia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fundacion Nacional de Dermatologia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ABF-BO-2016-102
Record Dates: First submitted 2017-03-09; First posted 2017-03-30 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2018-07

CONDITIONS: Leishmaniasis, Cutaneous; Leishmania Braziliensis Complex; Leishmaniasis, American; Leishmaniasis; American, Cutaneous
Keywords: leishmaniasis; L.braziliensis; paromomycin cream; intralesional pentamidine; leishmaniasis local therapy
MeSH Terms: conditions — Leishmaniasis, Cutaneous; Leishmaniasis, Mucocutaneous; Leishmaniasis | interventions — Paromomycin; Pentamidine

STUDY DESIGN:
Intervention Model Description: Patients will be randomized between Paromomycin cream applied topically once daily for 20 days (group 1--40 patients), pentamidine administered intralesionally at 120 ug/mm2 on days 1, 3, 5 (group 2-20 patients), and cream vehicle applied topically once daily for 20 days (group 3-20 patients).
Who Masked: Participant, Investigator
Masking Description: Group 1 (Paromomycin cream) will be compared to Group 3 (Vehicle cream). Both creams will have very similar physical characteristics and package. Group 2 (intralesional injection of pentamidine) will not be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 - Paromomycin cream (Experimental): 40 subjects will be included to receive 15% paromomycin in aquafilm base twice a day during 20 consecutive days. The lesion will be cleaned , then, a generous amount of the study drug (an amount sufficient to cover the area of the ulcer and the lesion border) will be applied to the lesion and rubbed into the ulcer using a gloved finger by a member of the clinical study staff. After application of the study drug, the patient will be observed for 15 minutes for signs of adverse events. If there are no signs of local toxicity, the area of the ulcer will be covered with extra study drug. For Days 2-20, the study drug will be applied and the lesion covered with a sterile gauze and tape dressing as on Day 1.
  Interventions: Drug: Paromomycin Sulfate
- Group 2. Local Injectable Pentamidine (Active Comparator): 20 subjects will be included to receive IL pentamidine [Pentacarinat® Sanofi-Aventis: 30 mg/ml] will administered at a dose of 120 ug (4 ul) per mm2 of lesion area 3 times (on days 1, 3, and 5) as per our previous experience.
  A small button of Xylocaine® will be applied by means of a thin needle at the four cardinal points of the lesion and then a small gauge (23g) needle will introduce the drug in each cardinal point. The needle will be moved in all directions to infiltrate of whole lesion and surrounding infiltrated area.
  Interventions: Drug: Pentamidine Isethionate
- Group 3. Vehicle control (Placebo Comparator): 10% Urea en parafilm cream will be used in similar ways as paromomycin cream in group 1
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Paromomycin Sulfate — topical application 2 times a day during 20 days
  Arms: Group 1 - Paromomycin cream
Drug: Pentamidine Isethionate — 3 Intralesional injections at days 1,3 and 5
  Arms: Group 2. Local Injectable Pentamidine
Other: Placebo — topical application 2 times a day during 20 days
  Arms: Group 3. Vehicle control

SUMMARY:
This protocol will compare topical paromomycin to standard intralesional (IL) antimony (Sb) to placebo for L braziliensis in Bolivia.

DETAILED DESCRIPTION:
Patients will be randomized between Paromomycin cream applied topically once daily for 20 days (group 1--40 patients), pentamidine administered intralesionally at 120 ug/mm2 on days 1, 3, 5 (group 2-20 patients), and cream vehicle applied topically once daily for 20 days (group 3-20 patients).

After treatment, all patients will be followed for 1, 3, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Gender: Male or female
* Age: >12 yrs of age
* Presentation: 1-to-2 ulcerative lesions, each < 30 mm in largest diameter and with a total lesion area <900 mm2.
* Parasitology: Parasitological confirmation of the lesion will be made by visualization or culture of Leishmania from the biopsy or aspirate of the lesion.

Exclusion Criteria:

* Previous treatment for leishmaniasis with Sb, pentamidine, amphotericin B, miltefosine, imidazoles, allopurinol in the last 3 months.
* Other diseases that would be likely in the PI's opinion to interact, either positively or negatively, with treatment.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2018-03-18 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Change of Lesion size | 6 months
  change of lesion area at 6 months after treatment compared to baseline

SECONDARY OUTCOMES:
Number of participants with treated-related adverse events | 1 month
  Adverse events will measured according to CTCAE 4.03

CONTACTS AND LOCATIONS:
Overall Officials: JAIME SOTO, MD, Principal Investigator — Fundacion Nacional de Dermatologia
Locations (2):
- Bolivia (2):
  - Hospital Local Palos Blancos, Palos Blancos, La Paz Department
  - Hospital Dermatologico de Jorochito, Jorochito, SC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oliveira-Neto MP, Schubach A, Mattos M, da Costa SC, Pirmez C. Intralesional therapy of American cutaneous leishmaniasis with pentavalent antimony in Rio de Janeiro, Brazil--an area of Leishmania (V.) braziliensis transmission. Int J Dermatol. 1997 Jun;36(6):463-8. doi: 10.1046/j.1365-4362.1997.00188.x. PMID 9248897
- [Background] Vasconcellos Ede C, Pimentel MI, Schubach Ade O, de Oliveira Rde V, Azeredo-Coutinho RB, Silva Fda C, Salgueiro Mde M, Moreira JS, Madeira Mde F, Baptista C, Valete-Rosalino CM. Intralesional meglumine antimoniate for treatment of cutaneous leishmaniasis patients with contraindication to systemic therapy from Rio de Janeiro (2000 to 2006). Am J Trop Med Hyg. 2012 Aug;87(2):257-60. doi: 10.4269/ajtmh.2012.11-0612. PMID 22855754
- [Background] Soto J, Rojas E, Guzman M, Verduguez A, Nena W, Maldonado M, Cruz M, Gracia L, Villarroel D, Alavi I, Toledo J, Berman J. Intralesional antimony for single lesions of bolivian cutaneous leishmaniasis. Clin Infect Dis. 2013 May;56(9):1255-60. doi: 10.1093/cid/cit049. Epub 2013 Feb 6. PMID 23390069
- [Background] Soto J, Paz D, Rivero D, Soto P, Quispe J, Toledo J, Berman J. Intralesional Pentamidine: A Novel Therapy for Single Lesions of Bolivian Cutaneous Leishmaniasis. Am J Trop Med Hyg. 2016 Apr;94(4):852-6. doi: 10.4269/ajtmh.15-0640. Epub 2016 Feb 22. PMID 26903605
- [Background] Ben Salah A, Ben Messaoud N, Guedri E, Zaatour A, Ben Alaya N, Bettaieb J, Gharbi A, Belhadj Hamida N, Boukthir A, Chlif S, Abdelhamid K, El Ahmadi Z, Louzir H, Mokni M, Morizot G, Buffet P, Smith PL, Kopydlowski KM, Kreishman-Deitrick M, Smith KS, Nielsen CJ, Ullman DR, Norwood JA, Thorne GD, McCarthy WF, Adams RC, Rice RM, Tang D, Berman J, Ransom J, Magill AJ, Grogl M. Topical paromomycin with or without gentamicin for cutaneous leishmaniasis. N Engl J Med. 2013 Feb 7;368(6):524-32. doi: 10.1056/NEJMoa1202657. PMID 23388004
- [Derived] Soto J, Soto P, Ajata A, Luque C, Tintaya C, Paz D, Rivero D, Berman J. Topical 15% Paromomycin-Aquaphilic for Bolivian Leishmania braziliensis Cutaneous Leishmaniasis: A Randomized, Placebo-controlled Trial. Clin Infect Dis. 2019 Feb 15;68(5):844-849. doi: 10.1093/cid/ciy619. PMID 30260376